CLINICAL TRIAL: NCT04866550
Title: Health in Smart Rurality: Impact on Coordination of Care of Telemonitoring and Data Centralization of Frailty Patients
Acronym: HIS2R
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-005-HIS2R
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Heart Failure
Keywords: Chronic diseases; Aging people; Cross-border care; New communication technology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Chronic Disease | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Connected tablet: Patients aged over 60, living at home, with heart failure and / or chronic obstructive pulmonary disease, potentially requiring care cross-border (France and Belgium).
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Daily record of temperature, weight, heart rate, systolic blood pressure and oxygen saturation

SUMMARY:
Chronic diseases are frequent (around 10% of the total population and 30% after 60 years) and accelerate age-related functional decline. Concerning cross-border patients, use of health services can be delayed given the distances, the lack of rapid road access and the limited availability of public transport and the complex organization of coordinated care.

One of the ways to reduce acute exacerbations and preserve the quality of life of patients is to detect warning signs early. One of the ways to do this is to use new communication technologies.

DETAILED DESCRIPTION:
The aim of the study is to assess feasibility of using a connected tablet to assess clinical parameters with an alert system in frailty patients aged over 60, living at home, with heart failure and / or chronic obstructive pulmonary disease, potentially requiring care cross-border (France and Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 60
* Patients living at home
* Patients with heart failure and / or chronic obstructive pulmonary disease,
* Patients potentially requiring care cross-border (France and Belgium).
* Patients agreeing to participate to the study

Exclusion Criteria:

* Patients who do not speak French
* Patients with severe cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 60, living at home, with heart failure and / or chronic obstructive pulmonary disease, potentially requiring care cross-border (France and Belgium).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Alert according to the connected tablet | 12 months
  significant change in temperature (egal or more 38°), weight (variation of more than 5%), heart rate (less than 50 beats per minute or greater than 100), systolic blood pressure (less than 85 mmHg or greater than 160 mmHg) and / or oxygen saturation (variation of more than 4%)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc NOVELLA, Principal Investigator — Université de Reims Champagne-Ardenne - CHU de Reims
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France